CLINICAL TRIAL: NCT06597422
Title: A Phase I, Single and Multiple Ascending-Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of STSP-0902 Ophthalmic Solution in Healthy Subjects
Brief Title: A Study of STSP-0902 Ophthalmic Solution in Healthy Subjects
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Staidson (Beijing) Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STSP-0902-02-001
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Neurotrophic Keratitis
Keywords: STSP-0902; Ophthalmic Solution; Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (10):
- Single Low Dose Arm (Experimental): Low dose of STSP-0902 ophthalmic solution to study eye. Single dose.
  Interventions: Drug: STSP-0902 ophthalmic solution
- Single Middle Dose Arm (Experimental): Middle dose of STSP-0902 ophthalmic solution to study eye. Single dose.
  Interventions: Drug: STSP-0902 ophthalmic solution
- Single High Dose Arm (Experimental): High dose of STSP-0902 ophthalmic solution to study eye. Single dose.
  Interventions: Drug: STSP-0902 ophthalmic solution
- Single Control Dose Arm (Experimental): STSP-0902 Placebo to study eye. Single dose.
  Interventions: Drug: STSP-0902 Placebo
- Multiple Low Dose Arm (Experimental): Low dose of STSP-0902 ophthalmic solution to study eye. Three times daily for a total of 8 days.
  Interventions: Drug: STSP-0902 ophthalmic solution
- Multiple Middle Dose Arm (Experimental): Middle dose of STSP-0902 ophthalmic solution to study eye. Three times daily for a total of 8 days.
  Interventions: Drug: STSP-0902 ophthalmic solution
- Multiple High Dose Arm (Experimental): High dose of STSP-0902 ophthalmic solution to study eye. Three times daily for a total of 8 days.
  Interventions: Drug: STSP-0902 ophthalmic solution
- Multiple Highest Dose Arm (Experimental): Middle dose of STSP-0902 ophthalmic solution to study eye. Six times daily for a total of 8 days.
  Interventions: Drug: STSP-0902 ophthalmic solution
- Multiple Control Dose Arm (Experimental): STSP-0902 Placebo to study eye. Multiple doses.
  Interventions: Drug: STSP-0902 Placebo
- Tear PK study Arm (Experimental): STSP-0902 ophthalmic solution to both eyes. Single dose.
  Interventions: Drug: STSP-0902 ophthalmic solution

INTERVENTIONS:
Drug: STSP-0902 ophthalmic solution — Eye drop, single dose
  Arms: Single High Dose Arm; Single Low Dose Arm; Single Middle Dose Arm
Drug: STSP-0902 Placebo — Eye drop, single dose
  Arms: Single Control Dose Arm
Drug: STSP-0902 ophthalmic solution — Eye drop, three times daily for a total of 8 days
  Arms: Multiple High Dose Arm; Multiple Low Dose Arm; Multiple Middle Dose Arm
Drug: STSP-0902 ophthalmic solution — Eye drop, six times daily for a total of 8 days
  Arms: Multiple Highest Dose Arm
Drug: STSP-0902 Placebo — Eye drop, multiple doses
  Arms: Multiple Control Dose Arm
Drug: STSP-0902 ophthalmic solution — Eye drop, single dose, tear samples will be collected
  Arms: Tear PK study Arm

SUMMARY:
This trial is a Phase I clinical study to evaluate the safety, tolerability, and pharmacokinetic (PK) characteristics of STSP-0902 ophthalmic solution in healthy subjects following single and multiple administrations. The study plans to enroll 80 healthy subjects and is divided into three stages: the single-dose study stage, the multiple-dose study stage, and the tear PK study stage. The single-dose and multiple-dose study stages are randomized, double-blind, placebo-controlled, dose-escalation designs, while the tear PK study stage is a single-dose, open-label design.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects aged between 18 and 45 years (inclusive).
2. Male subjects with a weight of ≥50.0 kg, and female subjects with a weight of ≥45.0 kg, with a Body Mass Index (BMI) between 19.0 and 26.0 kg/m² (inclusive).
3. Both eyes have a corrected visual acuity of ≥1.0, with normal or clinically insignificant results from eye examinations, including slit-lamp examination, intraocular pressure measurement, and fundus examination.
4. Schirmer I test results for both eyes are ≥10 mm/5 minutes (applicable only to subjects in the tear PK study stage).
5. Physical examination, vital signs, 12-lead ECG, chest imaging, and laboratory tests (including hematology, urinalysis, blood chemistry, and coagulation function) are normal or clinically insignificant during the screening period.
6. Subjects (including their partners) agree to use effective non-drug contraception during the trial and for 6 months after the last dose and must not plan to conceive, donate sperm, or donate eggs.
7. Subjects are fully informed about the content, process, and potential adverse effects of the trial, voluntarily sign the informed consent form, and be willing to complete the trial, follow-up, and related examinations according to the trial plan.

Exclusion Criteria:

1. History or current presence of any eye disease other than refractive errors (e.g., myopia, hyperopia, astigmatism).
2. History of any eye surgery (including laser correction surgery) or having only one functional eye.
3. Use of any topical eye medication (e.g., artificial tears, traditional Chinese medicine eye drops, antibiotic eye drops, recombinant monoclonal antibody eye drops, eye gels, etc.) within 1 month prior to screening.
4. Wearing contact lenses within 2 weeks before screening or needing to wear contact lenses during the clinical study.
5. Clinically significant abnormal results from corneal fluorescein staining (applicable only to subjects in the single-dose and multiple-dose study stages).
6. History or current presence of any severe systemic disease, including but not limited to cardiovascular, cerebrovascular, respiratory, gastrointestinal, endocrine, metabolic, neurological, hematological, oncological, immune, infectious, or psychiatric disorders, especially those that may affect the eyes (e.g., hypertension, diabetes, hyperthyroidism).
7. Abnormal and clinically significant results in any of the following tests: Hepatitis B surface antigen, Hepatitis C antibody, syphilis-specific antibody, or HIV test.
8. Allergy to any component of the investigational product or excipients, history of allergies (especially eye allergies), or a known history of food or drug allergies.
9. Vaccination within 1 month prior to screening or planned vaccination during the trial.
10. Use of prescription drugs, over-the-counter drugs, or herbal medicines within 2 weeks before screening.
11. History of treatment with nerve growth factor (NGF) drugs (e.g., murine NGF) or use of other neurotrophic drugs (e.g., B vitamins, fish oil, etc.) within 3 months before screening.
12. Underwent any major surgery within 6 months prior to screening or has plans for surgery during the trial.
13. History of smoking within 3 months before screening, defined as smoking more than 5 cigarettes or an equivalent amount of tobacco per day on average, or inability to abstain from any tobacco products during the study.
14. Regular alcohol consumption within 6 months before screening, defined as an average daily alcohol intake of more than 2 units (1 unit = 360 mL of beer, 45 mL of spirits with 40% alcohol, or 150 mL of wine), or a positive alcohol breath test result, or inability to abstain from any alcohol products during the study.
15. Daily consumption of more than 5 cups of coffee or strong tea (each cup ≥150 mL) within 3 months before screening, or inability to abstain during the study.
16. History of drug abuse (e.g., morphine, ketamine, tetrahydrocannabinol [cannabis], methamphetamine, MDMA [ecstasy], cocaine, etc.) or a positive drug abuse screening result.
17. Blood loss or blood donation >400 mL within 3 months prior to screening, or history of blood transfusion within 4 weeks before screening, or plans to donate blood or blood components during the trial or within 3 months after the trial ends.
18. Participation in any clinical trial and receipt of investigational drugs, devices, or vaccines within 3 months before screening.
19. Pregnant or lactating women, those with a positive blood pregnancy test, or women who have not used effective contraception within 2 weeks before screening.
20. Difficulty in administering eye drops, difficulty with venipuncture, inability to tolerate venipuncture for blood sampling, or history of needle phobia or blood phobia.
21. Any other condition that, in the investigator's opinion, makes the subject unsuitable for participation in this trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-20 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events related to study drug | Baseline to Day 28
  Number of participants with ocular and systemic adverse events as assessed by CTCAE v5.0.

SECONDARY OUTCOMES:
STSP-0902 concentration | Baseline to Day 28
  Measurement of STSP-0902 in plasma and tear after drug administration
Incidence of positive detection of anti-STSP-0902 antibodies | Baseline to Day 28
  Measurement of anti-drug antibody (ADA) to STSP-0902 in plasma after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Laichun Lu, Ph.D, Principal Investigator — Beijing Tongren Hospital
Locations (1):
- Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality, China